CLINICAL TRIAL: NCT01210638
Title: A Single Dose, Two-Period, Two-Treatment, Two-Sequence Crossover Bioequivalence Study of Oxymorphone Hydrochloride IR 10 mg Tablets, With a Naltrexone Block, Under Fasted Conditions
Brief Title: Bioequivalency Study of Oxymorphone Hydrochloride 10 mg Tablets Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OXYM-T10-PVFS-1
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Oxymorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxymorphone Hydrochloride (Active Comparator): Tablet
  Interventions: Drug: Oxymorphone
- Opana (Active Comparator): Tablet
  Interventions: Drug: Oxymorphone

INTERVENTIONS:
Drug: Oxymorphone — 10 mg tablet
  Other Names: Opana

SUMMARY:
The objective of this study was to prove the bioequivalence of Oxymorphone Hydrochloride 10 mg Tablets under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C. Treatment with known enzyme altering drugs. History of allergic or adverse response to oxymorphone hydrochloride or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Soran Hong, MD, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States